CLINICAL TRIAL: NCT05944614
Title: Towards Optimal Treatment of Marfan Syndrome
Acronym: TOWER
Status: Completed | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Netherlands Organisation for Scientific Research (Other Government)
Responsible Party: Principal Investigator, Dr. Ir. Pim van Ooij, Principal Investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: NL82669.018.22
Record Dates: First submitted 2023-06-28; First posted 2023-07-13 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Marfan Syndrome
Keywords: Magnetic Resonance Imaging; Aortic disease
MeSH Terms: conditions — Marfan Syndrome; Aortic Diseases | interventions — Magnetic Resonance Spectroscopy; Restraint, Physical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Aortic tissue acquired during aorta surgery
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Marfan Syndrome patients: Marfan Syndrome patients age 18-50 with a pathological FBN1 mutation
  Interventions: Other: Magnetic Resonance imaging (MRI) examination
- Healthy volunteers: Age and gender matched healthy control patients without a history of aortic disease.
  Interventions: Other: Magnetic Resonance imaging (MRI) examination

INTERVENTIONS:
Other: Magnetic Resonance imaging (MRI) examination — 3D CINE and 4 dimensional (4D) flow MRI sequence

SUMMARY:
The purpose of this study is to determine whether new magnetic resonance imaging techniques can be used as a biomarker of aortic disease severity in patients with Marfan syndrome.

ELIGIBILITY:
Inclusion Criteria:

* MFS patients with a known FBN1 mutation
* Between 18-50 years of age

Exclusion Criteria:

* Contraindication for MR imaging
* Mental retardation
* Pregnancy, or planned pregnancy during study period

Additional exclusion criteria healthy controls:

- History of aorta disease

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: All Marfan syndrome patients age 18-50 with a known FBN1 mutation are eligeble for participation. Only patients who are unable to undergo an MRI examination are excluded.
Sampling Method: Probability Sample
Enrollment: 148 (Actual)
Dates: Start 2023-02-23 (Actual); Primary Completion 2025-04-16 (Actual); Study Completion 2025-04-16 (Actual)

PRIMARY OUTCOMES:
Difference in 3D aortic displacement in millimeters between Marfan patients (MFS) and healthy volunteers. | Baseline
  aortic displacement in the thoracic aorta. normal values unknown, but single paper: Marfan patients range: 1.77 to 10.03 millimeters, volunteers 7.34 ± 1.69 millimeters. lower is worse.
Difference in pulse wave velocity, in meters per second between Marfan patients and healthy volunteers. | Baseline
  pulse wave velocity expressed in m/s in the thoracic aorta, normal values age dependent: but range +/- 4 - 30 m/s, higher is worse
Difference in oscillatory shear index (dimensionless) expressed in m/s between Marfan patients and healthy volunteers | Baseline
  oscillatory shear index (dimensionless) in the thoracic aorta, range between 0 - 0.5 (No normal values defined), higher is worse
Change in aortic displacement expressed in millimeters , between MFS patient aortas prior to compared to after PEARS procedure or conventional aortic surgery. | Change from baseline to 6 months after surgery
  aortic displacement expressed in millimeters in the thoracic aorta. Pre-post change unknown, however operated 3.60 +/- 1.0 millimeter versus native aorta 7.01 +/- 3.09 millimeters. Lower is worse
Change in aortic pulse wave velocity (meters/second), between MFS patient aortas prior to compared to after PEARS procedure or conventional aortic surgery. | Change from baseline to 6 months after surgery
  pulse wave velocity in the thoracic aorta expressed in meters/second. Higher is worse. normal values for change unknown.
Change in oscillatory shear index (dimensionless) between MFS patient aortas prior to compared to after PEARS procedure or conventional aortic surgery. | Change from baseline to 6 months after surgery
  oscillatory shear index (dimensionless) in the thoracic aorta. Higher is worse range between 0 -5.

SECONDARY OUTCOMES:
Difference in 3D aortic displacement expressed in mm between Marfan patients with and without a native aorta | Baseline
  aortic displacement in the thoracic aorta, lower is worse. operated 3.60 +/- 1.0 millimeter versus native aorta 7.01 +/- 3.09 millimeters
Difference in 3D aortic displacement expressed in mm between Marfan patients with aortic root diameter >4.5cm versus <4.5 cm | Baseline
  aortic displacement in the thoracic aorta, lower is worse. Normal values unknown.
Difference in 3D aortic displacement expressed in mm between Marfan patients with a haploinsufficient fibrillin 1 mutation versus dominant negative mutation | Baseline
  aortic displacement in the thoracic aorta. Lower is worse. Normal values unknown.
Difference in 3D aortic displacement expressed in mm between male versus female Marfan patients | Baseline
  aortic displacement in the thoracic aorta,Lower is worse. Normal values unknown.
Difference in 3D aortic displacement expressed in mm between Marfan patients based on antihypertensive medication used | Baseline
  aortic displacement in the thoracic aorta, Lower is worse. Normal values unknown.
Difference in pulse wave velocity, expressed in meters per second between Marfan patients with and without a native aorta | Baseline
  pulse wave velocity expressed in m/s in the thoracic aorta, Lower is worse. Normal values unknown. Single study in general aneurysm population: pre surgery: 18.0 +/-4.0 meters per second post surgery 20.6 +/- 6.0 meters per second. higher is worse
Difference in pulse wave velocity, expressed in m/s between Marfan patients with an aortic root diameter >4.5 cm versus <4.5 cm | Baseline
  pulse wave velocity expressed in m/s in the thoracic aorta. Higher is worse. Normal values unknown.
Difference in pulse wave velocity, expressed in m/s between Marfan patients with a haploinsufficient fibrillin-1 mutation versus a dominant negative mutation | Baseline
  pulse wave velocity expressed in m/s in the thoracic aorta. Higher is worse. Normal values unknown.
Difference in pulse wave velocity, expressed in m/s between male and female Marfan patients | Baseline
  pulse wave velocity expressed in m/s in the thoracic aorta Higher is worse. Normal values unknown.
Difference in pulse wave velocity, expressed in m/s between Marfan patients based on antihypertensive medication used | Baseline
  pulse wave velocity expressed in m/s in the thoracic aorta
Difference in oscillatory shear index (dimensionless) expressed in m/s between Marfan patients with and without a native aorta | Baseline
  oscillatory shear index (dimensionless) in the thoracic aorta. Higher is worse. Normal values unknown.
Difference in oscillatory shear index (dimensionless) expressed in m/s between Marfan patients with aortic root diameter >4.5cm versus <4.5 cm | Baseline
  oscillatory shear index (dimensionless) in the thoracic aorta. Higher is worse. Normal values unknown.
Difference in oscillatory shear index (dimensionless) expressed in m/s between Marfan patients with a haploinsufficient fibrillin 1 mutation versus dominant negative mutation | Baseline
  oscillatory shear index (dimensionless) in the thoracic aorta. Higher is worse. Normal values unknown.
Difference in oscillatory shear index (dimensionless) expressed in m/s between male versus female Marfan patients | Baseline
  oscillatory shear index (dimensionless) in the thoracic aorta. Higher is worse. Normal values unknown.
Difference in oscillatory shear index (dimensionless) expressed in m/s between Marfan patients based on antihypertensive medication used | Baseline
  oscillatory shear index (dimensionless) in the thoracic aorta. Higher is worse. Normal values unknown.
The correlation between regional wall shear stress and elastic fibre thickness in resected aorta tissue of MFS patients. | Baseline MRI with aortic surgery tissue
  Correlation of locally MRI measured wall shear stress and histologic findings in the thoracic aorta. Neither is worse. Normal values dependent on location of measurement, exploratory outcome. .

CONTACTS AND LOCATIONS:
Overall Officials: Pim Ooij, PhD, Principal Investigator — Amsterdam UMC
Locations (4):
- Netherlands (4):
  - Radboud University Medical Center, Nijmegen, Gelderland
  - Leiden University Medical Center, Leiden, North Holland
  - Amsterdam UMC, location AMC, Amsterdam
  - University Medical Center Groningen, Groningen

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared